CLINICAL TRIAL: NCT03104855
Title: Clearance of 25-hydroxyvitamin D in Cystic Fibrosis
Acronym: CF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Ian deBoer, Associate Professor, Medicine/Nephrology, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 50852; R01DK099199 (NIH); P30DK089507 (NIH)
Record Dates: First submitted 2017-02-17; First posted 2017-04-07 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-09

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; vitamin d catabolism
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single pharmacokinetics arm (Experimental)
  Interventions: Drug: d6-25-hydroxyvitamin D3

INTERVENTIONS:
Drug: d6-25-hydroxyvitamin D3 — intravenous administration of stable isotope-labeled D6-25(OH)D3

SUMMARY:
The goal of this study is to define 25(OH)D3 catabolism in CF patients using gold standard pharmacokinetics studies. Specifically, the investigators will evaluate the metabolic clearance of 25(OH)D3 among participants with CF and matched control subjects. The goal of this work is to provide the first comprehensive characterization of vitamin D metabolism in CF patients and promote novel hypotheses for subsequent studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Serum total 25(OH)D 10-50 ng/mL
* Diagnosis of cystic fibrosis in accordance with CF Foundation Guidelines; OR, normal CONTROL

Exclusion Criteria:

* Primary hyperparathyroidism
* Gastric bypass
* Tuberculosis or sarcoidosis
* Current pregnancy
* Child-Pugh Class B or C cirrhosis (i.e. cirrhosis with ascites, hepatic encephalopathy, bilirubin >=2 mg/dL, serum albumin <=3.5 g/dL, or PT >= 4 seconds)
* History of kidney transplantation or end stage renal disease treated with dialysis
* Use of vitamin D3 or vitamin D2 supplements exceeding a mean daily dose of 400 IU, within 3 months (wash-out allowed)
* Use of 1,25(OH)2D3 or an analogue, calcimimetics, or medications known to induce CYP24A1 within 4 weeks (wash-out allowed)
* Serum calcium > 10.1 mg/dL
* Hemoglobin < 9 g/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian de Boer, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- CF Group: Participants with cystic fibrosis
- Healthy Controls: Participants without cystic fibrosis
Period: Overall Study
Arm/Group | CF Group | Healthy Controls
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CF Group | Healthy Controls | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.3) | 24.8 (3.3) | 31.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Clearance of D6-25(OH)D3
Description: Metabolic clearance is calculated as the administered dose of 25(OH)D3 divided by the area under the plasma concentration-time curve (AUC). AUC is calculated using the linear trapezoidal method.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: mL/day
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
mL/day | 397 (73) | 342 (41)

2. Secondary Outcome: AUC of D6-25(OH)D3
Description: AUC is calculated using the linear trapezoidal method.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ng x day/mL
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
ng x day/mL | 58.3 (9.7) | 67.2 (8.3)

3. Secondary Outcome: Terminal Half-life of D6-25(OH)D3
Description: Terminal half-life is equal to ln2/k, where k is the slope of the terminal regression line estimated using ≥3 plasma concentrations.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: day
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
day | 16.2 (3.3) | 15.8 (1.6)

4. Secondary Outcome: Volume of Distribution of D6-25(OH)D3
Description: Volume of distribution in the central compartment is calculated as dose/C0, where dose is the administered dose of 25(OH)D3 and C0 is the initial (estimated) concentration of drug in plasma.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
Liters | 8.4 (1.4) | 7.2 (1.1)

5. Other Pre Specified Outcome: Metabolic Formation Clearance of D6-25(OH)D3 Metabolites
Description: Metabolic formation clearance is calculated as the daughter metabolite plasma AUC divided by the AUC of D6-25(OH)D3 (metabolite/parent AUC ratio). AUC is calculated using the linear trapezoidal method.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
ratio | 0.10 (0.02) | 0.08 (0.01)

6. Other Pre Specified Outcome: Serum Concentration of Calcium
Description: Change in the serum concentration of calcium from baseline to 7 days after 25(OH)D3
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
mg/dL | 0.00 (0.37) | 0.14 (0.27)

7. Other Pre Specified Outcome: Serum Concentration of Creatinine
Description: Change in the serum concentration of creatinine from baseline to 7 days after 25(OH)D3
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
mg/dL | 0.00 (0.03) | 0.00 (0.07)

8. Other Pre Specified Outcome: Serum Concentration of AST
Description: Change in the serum concentration of AST from baseline to 7 days after 25(OH)D3
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
Units/L | 0.60 (5.03) | -1.00 (2.55)

9. Other Pre Specified Outcome: Serum Concentration of ALT
Description: Change in the serum concentration of ALT from baseline to 7 days after 25(OH)D3
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: Units/L
Arm/Group | CF Group | Healthy Controls
Number analyzed (Participants) | 5 | 5
Units/L | 0.00 (0.00) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | CF Group | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/5 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CF Group (N=5) | Healthy Controls (N=5)
Pain or sensation in arm during infusion (General disorders) | 2 (2) | 0 (0)
Bruising after blood draw (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-30): https://cdn.clinicaltrials.gov/large-docs/55/NCT03104855/Prot_SAP_000.pdf